CLINICAL TRIAL: NCT02736227
Title: Biomarkers Predicting Successful Tacrolimus Withdrawal and Everolimus (Zortress) Monotherapy Early After Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Josh Levitsky, Associate Professor in Medicine-Gastroenterology and Hepatology and Surgery-Organ Transplantation, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00201794
Record Dates: First submitted 2016-03-24; First posted 2016-04-13 (Estimated); Results first posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Liver Transplantation
Keywords: liver transplantation; immunosuppression; everolimus; tacrolimus; kidney function; liver function; biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tacrolimus Withdrawal and Everolimus Monotherapy (Experimental): Tacrolimus will be tapered while continual use of everolimus.
  Interventions: Drug: Tacrolimus Withdrawal and Everolimus Monotherapy

INTERVENTIONS:
Drug: Tacrolimus Withdrawal and Everolimus Monotherapy — During the first month post-transplant, the subject receives everolimus (about 5-8 ng/mL) and tacrolimus with or without mycophenolic acid as part of standard of care procedures. At one month post-transplant, mycophenolic acid will be stopped and tacrolimus dosage will be reduced while continuing the dosage of everolimus. At three months post-transplant, tacrolimus dosage will be reduced by 50% of the daily dose each week. At four months post-transplant, tacrolimus will be discontinued.

SUMMARY:
Most patients who get a liver transplant must take immunosuppressants for the rest of their lives. However, this has occurred at the expense of chronic CNI toxicity, e.g. chronic kidney disease (CKD), metabolic complications, infections and malignancy. Everolimus (EVL) is a drug that may stabilize or improve kidney function for patients with chronic kidney disease (CKD) that has been caused by immunosuppressants. EVL is used for standard of care treatment to prevent transplant liver rejection in combination with other immunosuppressants, such as tacrolimus. The overall aim of this study is to examine a combination of two different immunosuppressants and EVL to determine if patients may have stabilized and/or improved kidney function without liver rejection. This study will look at how safe it is to slowly withdraw one anti-rejection medication while continuing to take the other medicine, and whether this can be done without liver rejection occurrence.

ELIGIBILITY:
Inclusion Criteria:

* Adult LT candidates ≥ 18 years of age
* Listed for or recent (within 1 month) recipient of deceased or living donor liver transplantation

Exclusion Criteria:

* Combined or previous organ transplantation
* Human immunodeficiency virus (HIV) infection
* Inability to provide informed consent or comply with the protocol.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-03; Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josh Levitsky, MD, MS, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Comprehensive Transplant Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From May 2016 to May 2018, 170 adult primary LT were performed at our center. 20 Subjects underwent tac (Tacrolimus)withdrwal.
  28 patients consented but 8 were removed
  Final sample for analysis is n=20
Pre-assignment Details: 28 patients consented but 8 were removed (n=1 withdrew, n=2 non compliant with protocol, n=2 new wound issues, n=1 high urine protein/creatinine ration and n=2 had neutropenia) Final sample for analysis is n=20
Groups:
- Graft Rejection After Tacrolimus Was Discontinued (REJ): Incidence of Acute Rejection after the initiation of Tacrolimus Withdrawl at Month 3 and 6
- No Graft Rejection After Tacrolimus Weaning (Non REJ): NON-REJ patients did not required liver biopsy during the trial
- Removed From Study Before Tac Withdrawl Started: Removed from study before Tac withdrawl started
Period: Overall Study
Arm/Group | Graft Rejection After Tacrolimus Was Discontinued (REJ) | No Graft Rejection After Tacrolimus Weaning (Non REJ) | Removed From Study Before Tac Withdrawl Started
Started | 5 | 15 | 8
Completed | 5 | 15 | 0
Not Completed | 0 | 0 | 8
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 5
Not completed — Non Compliant | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Withdrew From Study Before Tacrolimus Weaning: These subjects were removed after consenting. These subjects were not initiated on TAC weaning
- Total: Total of all reporting groups
Arm/Group | Graft Rejection After Tacrolimus Was Discontinued (REJ) | No Graft Rejection After Tacrolimus Weaning (Non REJ) | Withdrew From Study Before Tacrolimus Weaning | Total
Number analyzed (Participants) | 5 | 15 | 8 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (4.2) | 58.8 (6.8) | 56 (10.1) | 61.1 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 2 | 8
  Male | 4 | 10 | 6 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 5 | 15 | 8 | 28
Hepatocellular Carcinoma [Number; unit: participants] — Measure Analysis Population Description: Data was not collected for participant in the "Withdrew from study before Tacrolimus Weaning" Arm Population: no participants contributed data for the "Withdrew from study before Tacrolimus weaning"
  participants
    number analyzed (Participants) | 5 | 15 | 0 | 20
    (all) | 3 | 4 |  | 7
Primary Liver Disease- Hep C [Number; unit: participants] | 3 | 2 | 0 | 5
Primary Liver Disease- Alcohol [Number; unit: participants] | 1 | 5 | 0 | 6
Primary Liver Disease- Non Alcoholic Fatty Liver [Number; unit: participants] | 1 | 4 | 0 | 5
Primary Liver Disease- Other [Number; unit: participants] | 0 | 4 | 0 | 4
Tacrolimus Trough [Mean (Standard Deviation); unit: ng/ml] — Measure Description: Measure Analysis Population Description: Data was not collected for participant in the "Withdrew from study before Tacrolimus Weaning" Arm Population: Measure Analysis Population Description: no participants contributed data for the "Withdrew from study before Tacrolimus weaning"
  ng/ml
    number analyzed (Participants) | 5 | 15 | 0 | 20
    (all) | 5.4 (0.8) | 5.2 (1.4) |  | 5.2 (1.3)
Everolimus Trough [Mean (Standard Deviation); unit: ng/ml] — Population: Measure Analysis Population Description: no participants contributed data for the "Withdrew from study before Tacrolimus weaning"
  ng/ml
    number analyzed (Participants) | 5 | 15 | 0 | 20
    (all) | 5.3 (1.2) | 5.3 (2.3) |  | 5.3 (2.1)
Lab Value -White Blood Count [Mean (Standard Deviation); unit: 1000 *cells*/mm^3] — Population: Measure Analysis Population Description: no participants contributed data for the "Withdrew from study before Tacrolimus weaning"
  1000 *cells*/mm^3
    number analyzed (Participants) | 5 | 15 | 0 | 20
    (all) | 5.6 (1.9) | 3.7 (1.7) |  | 4.2 (1.9)
Lab Value -Hb [Mean (Standard Deviation); unit: g/dl] — Population: Measure Analysis Population Description: no participants contributed data for the "Withdrew from study before Tacrolimus weaning"
  g/dl
    number analyzed (Participants) | 5 | 15 | 0 | 20
    (all) | 11.9 (1.1) | 10.7 (2.5) |  | 11 (2.3)
Lab Value -Platelet count [Mean (Standard Deviation); unit: 1000 *cells*/mm^3] — Population: Measure Analysis Population Description: no participants contributed data for the "Withdrew from study before Tacrolimus weaning"
  1000 *cells*/mm^3
    number analyzed (Participants) | 5 | 15 | 0 | 20
    (all) | 144.6 (47.6) | 111.9 (59.2) |  | 119.7 (57.3)
Lab Value -eGFR-MDRD [Mean (Standard Deviation); unit: mL/min/1.73 m^2] — Population: Measure Analysis Population Description: no participants contributed data for the "Withdrew from study before Tacrolimus weaning"
  mL/min/1.73 m^2
    number analyzed (Participants) | 5 | 15 | 0 | 20
    (all) | 55.2 (15.6) | 60.3 (17.7) |  | 59 (17)
Lab Value -Total Bilirubin [Mean (Standard Deviation); unit: mg/dl] — Population: Measure Analysis Population Description: no participants contributed data for the "Withdrew from study before Tacrolimus weaning"
  mg/dl
    number analyzed (Participants) | 5 | 15 | 0 | 20
    (all) | 0.36 (0.1) | 0.8 (0.8) |  | 0.7 (0.7)
Lab Value -AST [Mean (Standard Deviation); unit: u/l] — Population: Measure Analysis Population Description: no participants contributed data for the "Withdrew from study before Tacrolimus weaning"
  u/l
    number analyzed (Participants) | 5 | 15 | 0 | 20
    (all) | 23.6 (5.4) | 15.4 (6.9) |  | 17.3 (7.4)
Lab Value -ALT [Mean (Standard Deviation); unit: u/l] — Population: Measure Analysis Population Description: no participants contributed data for the "Withdrew from study before Tacrolimus weaning"
  u/l
    number analyzed (Participants) | 5 | 15 | 0 | 20
    (all) | 28.2 (6.3) | 19.1 (7.3) |  | 21.3 (8)
Lab Value -Alk Phos [Mean (Standard Deviation); unit: u/l] — Population: Measure Analysis Population Description: no participants contributed data for the "Withdrew from study before Tacrolimus weaning"
  u/l
    number analyzed (Participants) | 5 | 15 | 0 | 20
    (all) | 95.2 (47.7) | 69.9 (24.6) |  | 75.9 (32.1)

OUTCOME MEASURES:

1. Primary Outcome: Amount of Treg Cells Observed in Peripheral Blood in Patients With and Without Rejection
Description: flow cytometry immunophenotyping and gene expression microassays to assess amount of Treg cells and mRNA in peripheral blood in patients with and without rejection (after Tacc withdrwal)
Time Frame: Six months post transplantation
Population: 15 patients did not reject and 5 had mild rejection responding to tacrolimus resumption.
Measure: Mean (Standard Deviation); unit: percentage of CD4 positive cell
Arm/Group | Graft Rejection After Tacrolimus Was Discontinued (REJ) | No Graft Rejection After Tacrolimus Weaning (Non REJ)
Number analyzed (Participants) | 5 | 15
percentage of CD4 positive cell | 10 (1) | 5 (.2)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Withdrew From Study Before Tacrolimus Weaning: Removed from study before Tac withdrawal started
Arm/Group | Graft Rejection After Tacrolimus Was Discontinued (REJ) | No Graft Rejection After Tacrolimus Weaning (Non REJ) | Withdrew From Study Before Tacrolimus Weaning
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/15 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/15 | 0/8
Other Adverse Events (participants affected / at risk) | 0/5 | 0/15 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT02736227/Prot_SAP_000.pdf